CLINICAL TRIAL: NCT04400890
Title: Randomized Double-Blind Placebo-Controlled Proof-of-Concept Trial of Resveratrol, a Plant Polyphenol, for the Outpatient Treatment of Mild Coronavirus Disease (COVID-19)
Brief Title: Randomized Proof-of-Concept Trial to Evaluate the Safety and Explore the Effectiveness of Resveratrol, a Plant Polyphenol, for COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Marvin McCreary, MD (Other)
Responsible Party: Sponsor-Investigator, Marvin McCreary, MD, Emergency Physician, Mount Carmel Health System
Organization: Mount Carmel Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: McCreary2020
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: Coronavirus; SARS-CoV-2; COVID; Vitamin D3; Cholecalciferol; Supplement; Polyphenol; Resveratrol; Stilbene; phytoalexin
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Resveratrol; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resveratrol with Vitamin D3 (Active Comparator): Resveratrol 1000mg four times per day for 15 days. Vitamin D3 100,000 IU on day 1
  Interventions: Drug: Resveratrol; Dietary Supplement: Vitamin D3
- Placebo with Vitamin D3 (Placebo Comparator): Placebo capsules 4 times per day for 15 days. Vitamin D3 100,000 IU on day 1
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Resveratrol — Resveratrol vs placebo given for 15 days.
  Other Names: Placebo
  Arms: Resveratrol with Vitamin D3
Dietary Supplement: Vitamin D3 — Vitamin D3 100,000 IU given on day one.

SUMMARY:
Resveratrol is a plant polyphenol (that is sold commercially as a supplement) that might help fight coronavirus as well as help protect the body from the effects of disease (COVID-19) caused by the infection. In this proof-of-concept pilot study we will compare the effects of resveratrol to placebo to assess the safety of the resveratrol and explore effectiveness.

DETAILED DESCRIPTION:
This randomized placebo-controlled trial is for the outpatient treatment of (Coronavirus Disease 2019) COVID-19. The purpose of this trial is to evaluate the safety and explore the effectiveness of resveratrol, a plant polyphenol, being re-purposed for patients with early COVID-19. Published in vitro data supports that this polyphenol inhibits coronavirus replication while separately published in silico (computer molecular docking analysis) reports have identified specific molecular targets of resveratrol against (Severe Acute Respiratory Syndrome - Coronavirus 2) SARS-CoV-2. Animal studies also demonstrate that resveratrol is effective at preventing lung injury and death in certain animal models of viral infections. Furthermore, the products long history as an anti-inflammatory might prevent the cytokine storm that is associated with worse outcomes in COVID-19.

200 subjects, 45 and older, (100 receiving the plant polyphenol, 100 receiving placebo) will be enrolled in study to compare whether taking resveratrol will reduce the rate of hospitalization. Subjects will take capsules 4 times a day for a minimum of 7 days (up to 15 days depending on duration of symptoms) plus both groups will receive Vitamin D3 100,000 IU to augment the effects of resveratrol. Resveratrol will be given as 1gm 4 times per day. Placebo tablets will contain brown rice flour in visually identical capsules. The primary outcome measure for this trial is reduction in hospitalization at 21 days from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who test positive for infection with SARS-CoV-2.
* Age ≥45 years
* Mild COVID-19 based on World Health Organization (WHO) Baseline Severity Categorization
* Symptom duration ≤ 10 days, or <72 hours of new respiratory symptoms.
* Patient must have access to the internet or a smartphone to complete surveys.
* English-speaking patients

Exclusion Criteria:

* Diagnosed or suspected cognitive impairment that would prevent the patient from cooperating with study procedures, as judged by the screening clinician
* Asymptomatic patients (e.g. patients who were screened without symptoms but tested positive)
* Known or suspected liver disease or Hepatitis C
* Known kidney disease with estimate Glomerular Filtration Rate (eGFR) <60
* Patients on warfarin, Novel Oral Anticoagulants (NOACs), HIV Protease Inhibitors, immunosuppressants, hydroxychloroquine/chloroquine, and other medication with a narrow therapeutic window.
* Allergy to grapes or rice.
* Co-morbidities with a high likelihood of hospitalization within 30 days (e.g., current cancer treatment, severe Chronic Obstructive Pulmonary Disease (COPD) or Congestive Heart Failure (CHF))
* Currently pregnant
* Hospitalization

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin R McCreary, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mt Carmel HealthSystems, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] McCreary MR, Schnell PM, Rhoda DA. Randomized double-blind placebo-controlled proof-of-concept trial of resveratrol for outpatient treatment of mild coronavirus disease (COVID-19). Sci Rep. 2022 Jun 29;12(1):10978. doi: 10.1038/s41598-022-13920-9. PMID 35768453
- [Derived] McCreary MR, Schnell PM, Rhoda DA. Randomized Double-blind Placebo-controlled Proof-of-concept Trial of Resveratrol for Outpatient Treatment of Mild Coronavirus Disease (COVID-19). Res Sq [Preprint]. 2021 Sep 13:rs.3.rs-861831. doi: 10.21203/rs.3.rs-861831/v1. PMID 34545357
- See also: Peer reviewed final publication — https://www.nature.com/articles/s41598-022-13920-9

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 13, 2020 and December 11, 2020, 1,694 patients were telephoned within 24-h of testing positive for COVID-19 to be recruited into the clinical trial . One-hundred-five were enrolled and randomized. Five withdrew after receiving treatment packets (four withdrew before starting treatment and one withdrew after one treatment day citing "too many pills" as reason for withdrawal).
Pre-assignment Details: One-hundred-five subjects were enrolled and randomized. Four participants withdrew before starting treatment. One participant withdrew after one treatment day citing "too many pills" as reason for withdrawal.
Groups:
- Resveratrol With Vitamin D3: Resveratrol 1000mg four times per day for up to 15 days (7 days minimum). Vitamin D3 100,000 IU on day 1
  Vitamin D3: Vitamin D3 100,000 IU given on day one.
- Placebo With Vitamin D3: Placebo capsules 4 times per day for up to 15 days (7 days minimum). Vitamin D3 100,000 IU on day 1
  Vitamin D3: Vitamin D3 100,000 IU given on day one.
Period: Overall Study
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Started (Intent-to-treat Population) | 53 | 52
Treated Per Protocol Population (Completed participation through 21-day primary outcome measures.) | 50 | 50
Completed | 50 | 50
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Between September 13, 2020 and December 11, 2020, 1,694 patients were telephoned within 24-h of testing positive for COVID-19 to be recruited into the clinical trial . One-hundred-five were enrolled and randomized. Five withdrew after receiving treatment packets (four withdrew before starting treatment and one withdrew after one treatment day citing "too many pills" as reason for withdrawal).
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3 | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (8.55) | 56.3 (9.46) | 56.0 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 24 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 43 | 45 | 88
  Unknown or Not Reported | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 47 | 46 | 93
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 1 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (4.68) | 31.4 (7.32) | 30.2 (6.2)
High Risk Comorbidity= YES [Count of Participants; unit: Participants] | 15 | 17 | 32
High Risk Comorbidity= NO [Count of Participants; unit: Participants] | 38 | 35 | 73
Chronic Lung Disease [Count of Participants; unit: Participants] | 10 | 9 | 19
Diabetes Mellitus [Count of Participants; unit: Participants] | 5 | 5 | 10
Cardiovascular Disease [Count of Participants; unit: Participants] | 3 | 3 | 6
Renal Disease [Count of Participants; unit: Participants] | 0 | 0 | 0
Liver Disease [Count of Participants; unit: Participants] | 0 | 0 | 0
Immunocompromised [Count of Participants; unit: Participants] | 0 | 0 | 0
Current Smoker [Count of Participants; unit: Participants] | 1 | 2 | 3
Former Smoker [Count of Participants; unit: Participants] | 8 | 12 | 20
Angiotensin Converting Enzyme Inhibitor (ACEI) / Angiotensin Receptor Blocker (ARB) use [Count of Participants; unit: Participants] | 5 | 10 | 15
Vitamin D use [Count of Participants; unit: Participants] | 6 | 2 | 8
Oral Steroid Use [Count of Participants; unit: Participants] | 2 | 2 | 4
Inhaled Steroid Use [Count of Participants; unit: Participants] | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization Rates for COVID-19
Description: Number of study participants admitted to the hospital within 21 days of randomization
Time Frame: 21 days from study randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Number analyzed (Participants) | 50 | 50
Participants | 1 | 3

2. Secondary Outcome: ICU Admission Rates
Description: Number of study participants admitted within 21 who subsequently get admitted to the ICU
Time Frame: 21 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

3. Secondary Outcome: Invasive Ventilation Rates
Description: Number of study participants who get admitted with 21 day of randomization who receiving invasive ventilation.
Time Frame: 21 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

4. Secondary Outcome: Pneumonia
Description: Number of study participants are diagnosed with pneumonia with 21 day of randomization
Time Frame: 21 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Number analyzed (Participants) | 50 | 50
Participants | 4 | 8

5. Secondary Outcome: Pulmonary Embolism
Description: Number of study participants are diagnosed with pulmonary embolism with 21 day of randomization
Time Frame: 21 days from start of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Number analyzed (Participants) | 50 | 50
Participants | 1 | 1

6. Secondary Outcome: Death
Description: Number of study participants who died with 21 day of randomization
Time Frame: Within 21 days from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

7. Other Pre Specified Outcome: Adverse Events
Description: Diarrhea, nausea, abdominal cramping
Time Frame: 60 days from randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: With 60 days of randomization
Arm/Group | Resveratrol With Vitamin D3 | Placebo With Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50 | 8/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol With Vitamin D3 (N=50) | Placebo With Vitamin D3 (N=50)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Resveratrol With Vitamin D3 (N=50) | Placebo With Vitamin D3 (N=50)
Increased Flatulence (Gastrointestinal disorders) | 20 | 16
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Hives (Skin and subcutaneous tissue disorders) | 5 | 2
Bruises easily (Skin and subcutaneous tissue disorders) | 3 | 5
Dry mouth (Gastrointestinal disorders) | 28 | 21
Sore Throat / Mount (Gastrointestinal disorders) | 18 | 17
Hoarse Voice (Respiratory, thoracic and mediastinal disorders) | 19 | 20
Problems Tasting / Smelling (Gastrointestinal disorders) | 30 | 24
Decreased Appetitis (Gastrointestinal disorders) | 29 | 26
Nausea (Gastrointestinal disorders) | 24 | 17
Vomiting (Gastrointestinal disorders) | 2 | 3
Heartburn (Gastrointestinal disorders) | 19 | 14
Bloating (Gastrointestinal disorders) | 27 | 19
Diarrhea (Gastrointestinal disorders) | 27 | 19
Constipation (Gastrointestinal disorders) | 14 | 14
Pain in Abdomen (Gastrointestinal disorders) | 19 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 31
Wheezing (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Racing Heartbeat (Cardiac disorders) | 16 | 19
Itchy Skin (Skin and subcutaneous tissue disorders) | 9 | 10
Dizziness (Nervous system disorders) | 22 | 16
Blurry Vision (Eye disorders) | 11 | 10
Redness or watery eyes (Eye disorders) | 16 | 16
Problems Concentrating (Nervous system disorders) | 19 | 21
Problems with memory (Nervous system disorders) | 14 | 12
Pain (General disorders) | 26 | 22
Headache (Nervous system disorders) | 31 | 30
Aching Muscle (Musculoskeletal and connective tissue disorders) | 26 | 24
Aching Joint (Musculoskeletal and connective tissue disorders) | 20 | 20
Nosebleeds (Blood and lymphatic system disorders) | 5 | 2
Shivering (General disorders) | 12 | 14

LIMITATIONS AND CAVEATS:
The actual rate of primary and secondary COVID-19 outcome measures were lower than expected. Therefore the study plan had inadequate number of participants and was therefore under-powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with SAP (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT04400890/Prot_SAP_001.pdf